CLINICAL TRIAL: NCT01092533
Title: Myfortic (Enteric-coated Mycophenolate Sodium) for the Treatment of Non-infectious Intermediate Uveitis - a Prospective, Controlled, Randomized Multicenter Trial
Brief Title: Myfortic for the Treatment of Non-infectious Intermediate Uveitis
Acronym: MYCUV-IIT02
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: STZ eyetrial (Other)
Collaborators: Novartis Pharmaceuticals (Industry); University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-009998-10
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Uveitis, Intermediate
MeSH Terms: conditions — Uveitis, Intermediate | interventions — Mycophenolic Acid; Prednisone; Prednisolone

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mycophenolate sodium + Prednisolone (Experimental): Mycophenolate sodium 1440 mg/day Prednisolone: initial dose 1 mg/kg/day, maintenance dose 5 mg/day
  Interventions: Drug: Myfortic; Drug: Decortin
- Prednisolone (Active Comparator): Prednisolone: initial dose 1 mg/kg/day, maintenance dose 5 mg/day
  Interventions: Drug: Decortin

INTERVENTIONS:
Drug: Myfortic — Myfortic 360 mg BID (during week 1) Myfortic 720 mg BID (from week 2 on) Maintenance dose Decortin 5mg/d
  Other Names: Mycophenolate Sodium
  Arms: Mycophenolate sodium + Prednisolone
Drug: Decortin — Maintenance dose 5 mg/d
  Other Names: Prednisolone

SUMMARY:
The objective of this clinical trial is to evaluate the efficacy, safety and tolerability of enteric-coated mycophenolate sodium (Myfortic®) in combination with low-dose corticosteroids (Decortin H®) compared to a monotherapy with low-dose corticosteroids (Decortin H®) in subjects with chronic intraocular inflammation (non-infectious intermediate uveitis).

DETAILED DESCRIPTION:
Mycophenolate mofetil (MMF), a pro-drug containing mycophenolic acid (MPA) as active agent, is approved for the treatment of acute graft rejection after kidney-, heart- and liver-transplantation, and was shown in 1995 to be effective in inhibiting the development of experimental autoimmune uveoretinitis. Further studies proved it to be a safe and effective steroid-sparing immunomodulatory for reducing the recurrence rate of non-infectious intermediate uveitis in humans. Although the adverse effect profile of MMF is comparatively benign, gastrointestinal adverse effects are a major concern and may limit its clinical benefit, because they may necessitate dose reduction, interruption, or even discontinuation of MMF.

An enteric-coated formulation of mycophenolate sodium (EC-MPS, Myfortic) has been developed especially to reduce MPA-related gastrointestinal adverse events. This clinical trial is a prospective controlled study to evaluate whether a Myfortic based regimen will be able to reduce the probability of a relapse compared to steroid therapy alone and to test whether a Myfortic based therapy provides a superior behaviour compared to a steroid regimen.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a documented at least 6 months history of unilateral or bilateral intermediate uveitis either idiopathic or due to non-infectious systemic disease (e.g. sarcoidosis, multiple sclerosis)
* Uveitis has to be considered to be active at the timepoint of enrolment according to at least one of the following criteria:

  * Grade 2+ or higher for vitreous haze
  * Grade 2+ or higher for anterior chamber cells
  * Presence of cystoid macular edema in OCT
  * Presence of retinal vessel leakage in FA
* Considered by the investigator to require systemic treatment.
* At least 18 years of age
* Not planning to undergo elective ocular surgery during the study
* Capable of understanding the purposes and risks of the study, able to give informed consent and to comply with the study requirements
* Subjects of both gender with reproductive potential who are sexually active agree to use contraception throughout the course of the study and for at least 3 months after completion of their study participation.
* Women of childbearing potential have to use a highly effective method of birth control defined as one which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly, such as implants, injectables, combined oral contraceptives, hormonal IUDs combined with barrier methods (e.g. condom, diaphragm or spermicide), sexual abstinence or vasectomised partner.
* Women of childbearing age must have a negative urine pregnancy test (UPT) within 48 hours prior to starting study drug and must not be lactating.

Female subjects of non-childbearing potential must meet at least one of the following criteria:

1. Postmenopausal females, defined as:

   c. Females over the age of 60 years. d. Females who are 45 to 60 years of age must be amenorrheic for at least 2 years.
2. Females who had a hysterectomy and/or bilateral oophorectomy.

Exclusion Criteria:

* Uveitis of infectious etiology
* Signs of tuberculosis in chest x-ray during the past 12 months before study entry
* Clinically suspected or confirmed central nervous system or ocular lymphoma
* Primary diagnosis of anterior or posterior uveitis
* Uncontrolled glaucoma or known steroid response
* Subjects who received treatment with a systemic immunosuppressive drug, a monoclonal antibody or any other biologic therapy within 90 days prior study entry
* Treatment with mycophenolate mofetil or mycophenolate sodium in the past
* Treatment with a periocular steroid injection within 6 weeks prior to study entry
* Presence of absolute contraindications for Decortin H and/or Myfortic as mentioned in the product informations (Appendix 1 and 2)
* Presence of relative contraindications for Decortin H and/or Myfortic as mentioned in the product information (Appendix 1 and 2) if the disorder leading to the relative contraindication can not sufficiently managed by concomitant medication.
* Recipients of a solid organ transplant
* Subjects with lens opacities or obscured ocular media upon enrolment making unable evaluation of the posterior eye segment
* Subjects with a history of herpes zoster or varicella infection within 3 months before enrollment
* Active, extraocular infection requiring the prolonged or chronic use of antimicrobial agents or the history/presence of active hepatitis A, B or C
* Seropositivity for human immunodeficiency virus (HIV)
* Alanine transaminase (ALT), aspartate transaminase (AST), or gamma-glutamyl transferase (GGT) ≥ 2x upper limit of normal (ULN)
* Severe anemia (hemoglobin < 8 g/dL), leukopenia (white blood cell count [WBC] < 2500 mm3), thrombocytopenia (platelet count < 80,000 mm3)
* Current malignancy or a history of malignancy within the previous 5 years
* Pregnant or lactating women
* Known allergy for fluorescein natrium
* Currently participating in another clinical trial with an investigational agent in the 30 days prior to study participation and/or has not recovered from any reversible effects or side effects of prior investigational agent
* Subjects with non-ocular, medically significant co-morbid conditions that impair normal activities, require systemic corticosteroids or immunosuppressives, or any medical condition that would likely have an impact on the participant´s ability to comply with the study visit schedule
* Any current or history of substance abuse, psychiatric disorder or a condition that, in the opinion of the investigator, may invalidate communication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-03; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Time from study entry to first relapse | 6 months
  A log-rank test will be used to evaluate differences between the treatment and control group with the null hypothesis of no differences in the survival distributions between the two groups and the alternative hypothesis of different survival distributions. A two-sided log-rank test will be used at a significance level of 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Deuter, Dr., Principal Investigator — Centre for Ophthalmology, University of Tuebingen
Locations (5):
- Germany (5):
  - Charité Universitätsmedizin Berlin, Augenklinik, Berlin
  - Universitäts-Augenklinik Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Heidelberg, Interdisziplinäres Uveitiszentrum, Heidelberg
  - Augenklinik der Ludwig-Maximilians-Universität München, München
  - Augenabteilung am St. Franziskus-Hospital Münster, Münster

REFERENCES:
- [Background] Jabs DA, Nussenblatt RB, Rosenbaum JT; Standardization of Uveitis Nomenclature (SUN) Working Group. Standardization of uveitis nomenclature for reporting clinical data. Results of the First International Workshop. Am J Ophthalmol. 2005 Sep;140(3):509-16. doi: 10.1016/j.ajo.2005.03.057. PMID 16196117
- [Background] Whitcup SM. Intermediate uveitis. In: Nussenblatt RB, Whitcup SM (eds.). Uveitis. Fundamentals and clinical practice. Elsevier publishers 2004: 291-300
- [Background] Chanaud NP 3rd, Vistica BP, Eugui E, Nussenblatt RB, Allison AC, Gery I. Inhibition of experimental autoimmune uveoretinitis by mycophenolate mofetil, an inhibitor of purine metabolism. Exp Eye Res. 1995 Oct;61(4):429-34. doi: 10.1016/s0014-4835(05)80138-1. PMID 8549684
- [Background] Zierhut M, Stubiger N, Aboalchamat W, Landenberger H, Bialasiewicz AA, Engelmann K. [Immunosuppressive therapy with mycophenolate mofetil (CellCept) in treatment of uveitis]. Ophthalmologe. 2001 Jul;98(7):647-51. doi: 10.1007/s003470170101. German. PMID 11490743
- [Background] Baltatzis S, Tufail F, Yu EN, Vredeveld CM, Foster CS. Mycophenolate mofetil as an immunomodulatory agent in the treatment of chronic ocular inflammatory disorders. Ophthalmology. 2003 May;110(5):1061-5. doi: 10.1016/S0161-6420(03)00092-7. PMID 12750115
- [Background] Lau CH, Comer M, Lightman S. Long-term efficacy of mycophenolate mofetil in the control of severe intraocular inflammation. Clin Exp Ophthalmol. 2003 Dec;31(6):487-91. doi: 10.1046/j.1442-9071.2003.00704.x. PMID 14641155
- [Background] Thorne JE, Jabs DA, Qazi FA, Nguyen QD, Kempen JH, Dunn JP. Mycophenolate mofetil therapy for inflammatory eye disease. Ophthalmology. 2005 Aug;112(8):1472-7. doi: 10.1016/j.ophtha.2005.02.020. PMID 16061096
- [Background] Siepmann K, Huber M, Stubiger N, Deuter C, Zierhut M. Mycophenolate mofetil is a highly effective and safe immunosuppressive agent for the treatment of uveitis : a retrospective analysis of 106 patients. Graefes Arch Clin Exp Ophthalmol. 2006 Jul;244(7):788-94. doi: 10.1007/s00417-005-0066-8. Epub 2005 Sep 15. PMID 16163494
- [Background] Mod A, Tamaska J, Adam E, Gidall J, Poros A, Kiraly A, Natonek K, Paloczi K, Hollan Z. [Importance of the detection of minimal residual disease in the management of acute leukemia]. Orv Hetil. 1991 Jun 16;132(24):1291-6, 1299. Hungarian. PMID 1857605
- [Background] Behrend M. Adverse gastrointestinal effects of mycophenolate mofetil: aetiology, incidence and management. Drug Saf. 2001;24(9):645-63. doi: 10.2165/00002018-200124090-00002. PMID 11522119
- [Background] Budde K, Curtis J, Knoll G, Chan L, Neumayer HH, Seifu Y, Hall M; ERL B302 Study Group. Enteric-coated mycophenolate sodium can be safely administered in maintenance renal transplant patients: results of a 1-year study. Am J Transplant. 2004 Feb;4(2):237-43. doi: 10.1046/j.1600-6143.2003.00321.x. PMID 14974945
- [Background] Hachinski VC, Wilson JX, Smith KE, Cechetto DF. Effect of age on autonomic and cardiac responses in a rat stroke model. Arch Neurol. 1992 Jul;49(7):690-6. doi: 10.1001/archneur.1992.00530310032009. PMID 1497494
- [Background] Pleyer U, Ruokonen P, Schmidt N, Feist E, Hohne M, Stanojlovic S. [Mycophenol acid in ocular automimmune disorders--can we optimise this therapy?]. Klin Monbl Augenheilkd. 2008 Jan;225(1):66-9. doi: 10.1055/s-2008-1027134. German. PMID 18236373